CLINICAL TRIAL: NCT02853981
Title: Clamp-crush Technique Versus Harmonic Scalpel in Living Donor Hepatectomy. A Single Blinded Randomized Controlled Trial
Brief Title: Clamp-crush Technique Versus Harmonic Scalpel in Living Donor Hepatectomy
Acronym: KK_HS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmad Mohammad Ahmad Sultan, Assistant professor of general surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GEC_LTx_Surg_216
Record Dates: First submitted 2016-03-11; First posted 2016-08-03 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Hepatic Transplantation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Harmonic scalpel group (Active Comparator): group of donors whom will undergo liver transection using harmonic scalpel.
  Interventions: Device: Harmonic scalpel
- clamp-crush group (Active Comparator): group of donors whom will undergo liver transection using Kelly clamp.
  Interventions: Device: Kelly clamp crush technique

INTERVENTIONS:
Device: Harmonic scalpel — a method for liver parenchymal transection
  Arms: Harmonic scalpel group
Device: Kelly clamp crush technique — a method for liver parenchymal transection
  Arms: clamp-crush group

SUMMARY:
The purpose of this study is to determine whether clamp-crush technique for liver parenchymal transection is as safe as Harmonic scalpel device. outcomes will include: perioperative mortality, surgery-related complications, blood loss, amount of blood loss during hepatectomy, operating time, transection speed, markers of liver parenchymal injury and hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Liver right lobe donors

Exclusion Criteria:

-

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
blood loss during hepatectomy | intraoperative
  bleeding during transection phase will be calculated in mL. based on the blood in the sucker machine and the surgical towels

SECONDARY OUTCOMES:
transection speed | intraoperative
  the transection speed will be calculated in minutes based on the relation between the transecition time divided by the surface area of the raw area of the graft measured on the backtable.
liver pathology from the cut margin | intraoperative
  the area of necrosis will be measured in millimeters by the pathologist

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad M Sultan, MD, Study Director — Assistant prof of general surgery
Locations (1):
- Gastro-enterolgy surgical center, Mansoura University, Al Mansurah, Al-Dakahleia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sultan AM, Shehta A, Salah T, Elshoubary M, Elghawalby AN, Said R, Elmorshedi M, Marwan A, Shiha U, Fathy O, Wahab MA. Clamp-Crush Technique Versus Harmonic Scalpel for Hepatic Parenchymal Transection in Living Donor Hepatectomy: a Randomized Controlled Trial. J Gastrointest Surg. 2019 Aug;23(8):1568-1577. doi: 10.1007/s11605-019-04103-5. Epub 2019 Jan 22. PMID 30671805